CLINICAL TRIAL: NCT04966000
Title: Development of a Neuroimaging Biomarker to Identify Optimal Candidates for Prism Adaptation Treatment
Brief Title: Neurobiomarker for Prism Adaptation Treatment Response
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no time to complete study in this format
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00140741
Record Dates: First submitted 2021-06-30; First posted 2021-07-16 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2023-09

CONDITIONS: Perceptual Disorders; Stroke; Biomarker
Keywords: stroke; Prism Adaptation Therapy; spatial neglect
MeSH Terms: conditions — Perceptual Disorders; Stroke

STUDY DESIGN:
Intervention Model Description: a single group pre-post pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prism Adaptation Therapy (Experimental): 10 sessions (60 trials each) 1x/day of Prism Adaptation Therapy
  Interventions: Behavioral: Prism Adaptation Therapy

INTERVENTIONS:
Behavioral: Prism Adaptation Therapy — Participants wear goggles with built-in prisms (a 20-diopter lens) that shift the visual scene to the right. While wearing the googles they reach to and cross out 60 lines/circles, requiring them to learn to reach more leftward than the visual targets appear. Participants can only see the end of their movements.
  Other Names: PAT

SUMMARY:
Preliminary data will be collected about which individuals with spatial neglect from right hemisphere stroke (aiming vs perceptual neglect) improve with Prism Adaptation Training and if there is a particular pattern of damage in the brain that predicts both the type of neglect experienced and whether neglect is improved following Prism Adaptation Training

DETAILED DESCRIPTION:
For preliminary data, twelve individuals with right hemisphere stroke and spatial neglect will participate. After pretesting for type of neglect and its severity, they will have an MRI with Diffusion Tensor Imaging (DTI). Then they will complete 10 sessions of Prism Adaptation Therapy and complete neglect post-testing. Response to Prism Adaptation Therapy will be assessed by comparing neglect scores pre- and post-training. Traditional lesion mapping, structural and functional lesion disconnectivity analyses, and tract-based spatial statistics of DTI measures will be used to examine whether any patterns of damage/dysfunction are related to a diagnosis of aiming neglect and response to Prism Adaptation Therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1) within 1 month of right hemisphere stroke

  2) suspected of having unilateral spatial neglect

  3) able to provide consent

  4) likely to remain in rehabilitation for 10-12 days or willing to return to the University to complete 10 sessions of treatment and post-treatment testing

  5) able to have an MRI

  6) will be or has been admitted to the Craig H. Neilson Rehabilitation Hospital for rehabilitation or is able to come to the Craig H. Neilson Rehabilitation Hospital for prism adaptation therapy sessions.

  7) age 18-90 years

  8) able to sit in a wheelchair or other chair for 1 hour

  9) able to point straight ahead and hold a pen with right hand

Exclusion Criteria:

* 1) other neurologic, medical that would interfere with ability to complete the testing or training

  2) no uncorrected visual or hearing problems, other than hemianopsia

  3) contraindications to MRI

  4) unable to provide consent due to significant aphasia or cognitive impairment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Catherine Bergego Scale | baseline before prism adaptation therapy
  asks the impact of neglect behavior on 20 everyday tasks using a 0-3 rating scale. Higher scores = more neglect impact. Total score is sum of item scores
Catherine Bergego Scale | post-intervention immediately after prism adaptation therapy
  asks the impact of neglect behavior on 20 everyday tasks using a 0-3 rating scale. Higher scores = more neglect impact. Total score is sum of item scores

SECONDARY OUTCOMES:
Behavioral Attention Test conventional subtests | baseline pre-prism adaptation therapy
  traditional neuropsychological subtests (line crossing, letter cancelation, star cancellation, figure and shape copying, line bisection, and representational drawing). Total score is the sum of scores on subtests with highest score being 146. A score of 129 or higher indicates neglect
Behavioral Attention Test conventional subtests | post-intervention immediately after prism adaptation therapy
  traditional neuropsychological subtests (line crossing, letter cancelation, star cancellation, figure and shape copying, line bisection, and representational drawing). Total score is the sum of scores on subtests with highest score being 146. A score of 129 or higher indicates neglect

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided
We may share data with colleagues at Emory University and Washington University as they are engaged in similar research and combining data may allow for greater statistical power.

REFERENCES:
- [Result] Goedert KM, Chen P, Boston RC, Foundas AL, Barrett AM. Presence of Motor-Intentional Aiming Deficit Predicts Functional Improvement of Spatial Neglect With Prism Adaptation. Neurorehabil Neural Repair. 2014 Jun;28(5):483-93. doi: 10.1177/1545968313516872. Epub 2013 Dec 27. PMID 24376064
- [Result] Goedert KM, Chen P, Foundas AL, Barrett AM. Frontal lesions predict response to prism adaptation treatment in spatial neglect: A randomised controlled study. Neuropsychol Rehabil. 2020 Jan;30(1):32-53. doi: 10.1080/09602011.2018.1448287. Epub 2018 Mar 20. PMID 29558241